CLINICAL TRIAL: NCT01147276
Title: Study of the Effect of Vildagliptin on Glucagon Counterregulation Response During Hypoglycemia in Patients With Type 1 Diabetes
Brief Title: Vildagliptin and the Glucagon Response to Hypoglycemia in Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bo Ahren, Professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Lund University Diabetes 002
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes; Hypoglycemia
Keywords: DPP-4; GLP-1; Glucagon; Catecholamines; Counterregulation; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vildagliptin (Experimental): Vildagliptin (50 mg BID) given for four weeks
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin (50 mg BID) in four weeks
  Other Names: Galvus

SUMMARY:
The study examines whether DPP-4 inhibition by vildagliptin affects the glucagon counterregulatory response to hypoglycemia in type 1 diabetes.

DETAILED DESCRIPTION:
Vildagliptin (50 mg BID) or placebo is given as add-on to insulin treatment for four weeks in patients with type 1 diabetes. Then, a hypoglycemic clamp (2.5 mmol/l glucose) is undertaken with the determination of glucagon.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Age >18 years
* HbA1c 6.5-8,5%

Exclusion Criteria:

* Pregnancy
* Lactation
* Acute infection
* Liver disease
* Treatment with cortisol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Glucagon response to hypoglycemia | 45 min
  Change in glucagon from before hypoglycemic clamp until after 45 min

SECONDARY OUTCOMES:
Catecholamine response to hypoglycemic | 45 min
  Change in catecholamines from before hypolycemic clamp to 45 min

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ahrén, PhD MD, Principal Investigator — Lund University
Locations (1):
- Department of Clinical Sciences Lund, Lund University, Lund, Sweden

REFERENCES:
- [Derived] Farngren J, Persson M, Schweizer A, Foley JE, Ahren B. Vildagliptin reduces glucagon during hyperglycemia and sustains glucagon counterregulation during hypoglycemia in type 1 diabetes. J Clin Endocrinol Metab. 2012 Oct;97(10):3799-806. doi: 10.1210/jc.2012-2332. Epub 2012 Aug 1. PMID 22855332